CLINICAL TRIAL: NCT02811965
Title: Evaluation of Heel Offloading Devices for Reducing Heel Contact Pressures in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeRoyal Industries, Inc. (Industry)
Collaborators: Lincoln Memorial University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 534
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Heel Pressure Ulceration Prevention Strategies
Keywords: heel; pressure ulcer; pressure mapping
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Each research subject will have pressure mapping performed on his or her right foot in the 7 conditions described for each study arm to determine the contact forces experienced by the heel in each off-loading condition. Each intervention will be randomly applied.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Control (No Intervention): Pressure mapping is performed without a heel offloading intervention applied.
- Pillow Condition 1 (Experimental): Pressure mapping is performed with the Pillow condition 1 intervention applied to the heel.
  Interventions: Other: Pillow Condition 1
- Pillow Condition 2 (Experimental): Pressure mapping is performed with the Pillow condition 2 applied to the heel.
  Interventions: Other: Pillow Condition 2
- Heel Foam Pillow (Experimental): Pressure mapping is performed with the heel foam pillow device applied to the heel.
  Interventions: Device: Heel Foam Pillow
- Offloading Device A (Experimental): Pressure mapping is performed with Offloading Device A applied to the heel.
  Interventions: Device: Offloading Device A
- Offloading Device B (Experimental): Pressure mapping is performed with Offloading Device B applied to the heel.
  Interventions: Device: Offloading Device B
- Offloading Device C (Experimental): Pressure mapping is performed with Offloading Device C applied to the heel.
  Interventions: Device: Offloading Device C

INTERVENTIONS:
Other: Pillow Condition 1 — The heel is offloaded by placing the heel on a standard hospital pillow.
  Arms: Pillow Condition 1
Other: Pillow Condition 2 — The heel is offloaded by placing a standard hospital pillow under the calf suspending the heel above the hospital bed mattress.
  Arms: Pillow Condition 2
Device: Heel Foam Pillow — An economy heel offloading device constructed of egg shell foam.
  Arms: Heel Foam Pillow
Device: Offloading Device A — Heel offloading device that utilizes open cell foam to offload the heel. Device has a published clinical study demonstrating effectiveness at reducing heel ulceration rate.
  Arms: Offloading Device A
Device: Offloading Device B — Heel offloading device that utilizes pressure absorbing filling to offload the heel. Device has a published clinical study demonstrating effectiveness at reducing heel ulceration rate
  Arms: Offloading Device B
Device: Offloading Device C — Heel offloading device that utilizes a similar pressure absorbing filling to Offloading Device B; however this device does not have published clinical literature demonstrating effectiveness at reducing heel ulceration in the clinic.
  Other Names: PRUventor® Heel Off-loading Device
  Arms: Offloading Device C

SUMMARY:
Prevention of heel pressure ulceration is a major clinical concern. Clinical research has shown that heel-offloading devices are effective at preventing heel ulceration when compared to no offloading or sub-optimal offloading methods (i.e. use of a hospital pillow to offload the heel). As a result, a plethora of heel-offloading devices have been developed that utilize different designs and materials to offload the heel. Despite the availability of these devices, some healthcare facilities still employ no heel offloading or utilize sub-optimal heel offloading strategies. It is also difficult for clinicians to compare the effectiveness of different heel offloading device without conducting extensive clinical evaluations. Pressure mapping of the pressure experienced by the heel while offloaded offers a potential method to assess the effectiveness of different heel offloading strategies.

The primary hypothesis of this study is that the three tested heel offloading devices will significantly decrease the heel contact forces compared to no offloading and sub-optimal heel offloading conditions. The secondary objective is to quantify differences in heel contact forces experienced by the heel when placed in each heel offloading device to demonstrate the utility of pressure mapping as a tool to evaluate the effectiveness of different heel offloading devices.

The study will recruit 21 healthy volunteers as research subjects with 7 having a normal BMI, 7 having an overweight BMI, and 7 having an obese BMI. Pressure mapping will be conducted on each research subject for seven randomly applied conditions while the patient lies comfortably in a hospital bed. The seven conditions include no heel offloading, 3 sub-optimal offloading conditions, and offloading in 3 different heel-offloading devices. Pressure measurements corresponding to the heel will be used to determine the average peak pressure contact force for each research subject in each condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* No musculoskeletal injury in the past month
* Body Mass Index (BMI) between 18.5 and 39.9

Exclusion Criteria:

* 17 years old or younger
* Musculoskeletal injury in the past month
* Pregnant or lactating female
* History of heel pressure ulceration
* BMI below 18.5 or above 39.9

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Savage, DNP, Principal Investigator — Lincoln Memorial University
Locations (1):
- Lincoln Memorial University; Cedar Bluff Campus, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Research Subjects: Each research subject will have pressure mapping performed on his or her right foot in the 7 interventions listed to determine the contact forces experienced by the heel in each off-loading condition. Each intervention will be randomly applied.
Period: Overall Study
Arm/Group | Healthy Research Subjects
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Research Subjects
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight, Continuous [Mean (Standard Deviation); unit: lbs] | 168.6 (43.5)
Height, Continuous [Mean (Standard Deviation); unit: inches] | 65.7 (4.2)
Body Mass Index (BMI), Continuous [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (5.7)
BMI, Categorical [Count of Participants; unit: Participants]
  18.5 < BMI < 24.9 | 8
  25 < BMI < 29.9 | 7
  30 < BMI | 6

OUTCOME MEASURES:

1. Primary Outcome: Average Contact Force Exerted on the Heel
Description: Average contact force calculated from an area of 40.32 cm^2 that encompassed the entire posterior heel. Pressure readings obtained by pressure mapping
Time Frame: 5 minutes of pressure mapping
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Pillow Condition 1 | Pillow Condition 2 | Heel Foam Pillow | Offloading Device A | Offloading Device B | Offloading Device C
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 21 | 21 | 21
mmHg | 60.25 (13.68) | 39.74 (10.84) | 5.57 (3.94) | 29.34 (7.67) | 24.50 (9.63) | 20.72 (10.25) | 7.00 (12.51)
Statistical Analysis 1: Comparison: Control vs Pillow Condition 1 vs Pillow Condition 2 vs Heel Foam Pillow vs Offloading Device A vs Offloading Device B vs Offloading Device C; Test type: Superiority; p < 0.00005, Repeated Measures ANOVA — A priori threshold p < 0.05
Statistical Analysis 2: Comparison: Control vs Pillow Condition 1; Test type: Superiority; p = 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 3: Comparison: Control vs Pillow Condition 2; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 4: Comparison: Control vs Heel Foam Pillow; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 5: Comparison: Control vs Offloading Device A; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 6: Comparison: Control vs Offloading Device B; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 7: Comparison: Control vs Offloading Device C; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 8: Comparison: Pillow Condition 1 vs Pillow Condition 2; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 9: Comparison: Pillow Condition 1 vs Heel Foam Pillow; Test type: Superiority; p = 0.01, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 10: Comparison: Pillow Condition 1 vs Offloading Device A; Test type: Superiority; p = 0.0002, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 11: Comparison: Pillow Condition 1 vs Offloading Device B; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 12: Comparison: Pillow Condition 1 vs Offloading Device C; Test type: Superiority; p < 0.00005, t-test, 2 sided
Statistical Analysis 13: Comparison: Pillow Condition 2 vs Heel Foam Pillow; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 14: Comparison: Pillow Condition 2 vs Offloading Device A; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 15: Comparison: Pillow Condition 2 vs Offloading Device B; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 16: Comparison: Pillow Condition 2 vs Offloading Device C; Test type: Superiority; p = 0.24, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 17: Comparison: Heel Foam Pillow vs Offloading Device A; Test type: Superiority; p = 0.14, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 18: Comparison: Heel Foam Pillow vs Offloading Device B; Test type: Superiority; p = 0.0093, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 19: Comparison: Heel Foam Pillow vs Offloading Device C; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 20: Comparison: Offloading Device A vs Offloading Device B; Test type: Superiority; p = 0.14, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 21: Comparison: Offloading Device A vs Offloading Device C; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 22: Comparison: Offloading Device B vs Offloading Device C; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05

2. Primary Outcome: Peak Pressure Index on the Heel
Description: Peak pressure index calculated by centering a 3 X 3 region of interest (14.52 cm^2) over maximum pressure sensor reading within the region of interest encompassing the heel.
Time Frame: 5 minutes of pressure mapping
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | Pillow Condition 1 | Pillow Condition 2 | Heel Foam Pillow | Offloading Device A | Offloading Device B | Offloading Device C
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 21 | 21 | 21
mmHg | 120.15 (23.88) | 69.93 (17.63) | 10.97 (8.42) | 48.06 (9.87) | 39.88 (18.01) | 32.18 (14.71) | 12.51 (8.26)
Statistical Analysis 1: Comparison: Control vs Pillow Condition 1 vs Pillow Condition 2 vs Heel Foam Pillow vs Offloading Device A vs Offloading Device B vs Offloading Device C; Test type: Superiority; p < 0.00005, Repeated Measures ANOVA — A priori threshold p<0.05
Statistical Analysis 2: Comparison: Control vs Pillow Condition 1; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 3: Comparison: Control vs Pillow Condition 2; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 4: Comparison: Control vs Heel Foam Pillow; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 5: Comparison: Control vs Offloading Device A; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 6: Comparison: Control vs Offloading Device B; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 7: Comparison: Control vs Offloading Device C; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 8: Comparison: Pillow Condition 1 vs Pillow Condition 2; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 9: Comparison: Pillow Condition 1 vs Heel Foam Pillow; Test type: Superiority; p = 0.0011, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 10: Comparison: Pillow Condition 1 vs Offloading Device A; Test type: Superiority; p = 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 11: Comparison: Pillow Condition 1 vs Offloading Device B; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 12: Comparison: Pillow Condition 1 vs Offloading Device C; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 13: Comparison: Pillow Condition 2 vs Heel Foam Pillow; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 14: Comparison: Pillow Condition 2 vs Offloading Device A; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 15: Comparison: Pillow Condition 2 vs Offloading Device B; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 16: Comparison: Pillow Condition 2 vs Offloading Device C; Test type: Superiority; p = 0.53, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 17: Comparison: Heel Foam Pillow vs Offloading Device A; Test type: Superiority; p = 0.092, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 18: Comparison: Heel Foam Pillow vs Offloading Device B; Test type: Superiority; p = 0.0044, t-test, 2 sided
Statistical Analysis 19: Comparison: Heel Foam Pillow vs Offloading Device C; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 20: Comparison: Offloading Device A vs Offloading Device B; Test type: Superiority; p = 0.084, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 21: Comparison: Offloading Device A vs Offloading Device C; Test type: Superiority; p < 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05
Statistical Analysis 22: Comparison: Offloading Device B vs Offloading Device C; Test type: Superiority; p = 0.00005, t-test, 2 sided — P-value adjusted with Holm-Bonferroni Correction for multiple comparison. A priori threshold p<0.05

ADVERSE EVENTS:
Arm/Group | Control | Pillow Condition 1 | Pillow Condition 2 | Heel Foam Pillow | Offloading Device A | Offloading Device B | Offloading Device C
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21 | 0/21 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less